CLINICAL TRIAL: NCT06405152
Title: Assessment of Macrophage Activation syndromE in STill's Disease: Retrospective Chart Analysis of Patient HistorY, Symptom Resolution and Treatment Characteristics
Brief Title: Assessment of Macrophage Activation syndromE in STill's Disease
Acronym: AMETHYST
Status: Completed | Type: Observational
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Other Study IDs: Sobi.Emapalumab-105
Record Dates: First submitted 2024-04-09; First posted 2024-05-08 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Macrophage Activation Syndrome; Still's Disease, Adult-Onset; Stills Disease, Juvenile-Onset
MeSH Terms: conditions — Macrophage Activation Syndrome; Still's Disease, Adult-Onset; Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Other: Chart review — Retrospective Chart Review

SUMMARY:
Assessment of Macrophage activation syndrome in STill's disease: retrospective chart analysis of patient History, Symptom resolution and Treatment characteristics

DETAILED DESCRIPTION:
This is an observational, retrospective cohort study on the treatment utilization and outcomes of Macrophage Activation Syndrome (MAS) refractory to glucocorticoids (GC) in patients with Still's disease. The study will be conducted entirely through medical chart abstraction; all data will be taken from the patient's medical record, with no additional assessments.

ELIGIBILITY:
Inclusion Criteria:

* Age >6 months and ≤80 years at the beginning of the index MAS episode.
* Diagnosis of Still's disease (sJIA (systemic Juvenile Idiopathic Arthritis) or AOSD (Adult Onset Stills Disease) diagnosis).
* Diagnosis of MAS according to treating physician in the medical record.
* Patients who have received at least 3 consecutive days of GC after diagnosis of MAS and/or are judged by the Investigator to be refractory to GC due to clinical worsening of patient's condition .
* The onset of the index MAS episode occurred between 01 January 2012 and 30 September 2022.

Exclusion Criteria:

* A diagnosis of primary Hemophagocytic Lymphohistiocytosis (HLH) prior to the beginning of the index MAS episode.
* Confirmed malignancy prior to the beginning of the index MAS episode.
* Patient treated with any investigational product as a part of clinical trial during the index MAS episode.

Ages: 6 Months to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include patients with Still's disease who were diagnosed with MAS that was refractory to GC treatment.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year
  The proportion of patients alive after 1-year of follow-up
Time to laboratory value normalization | From Index date up to 26 weeks
  Time to normalization for the key laboratory values
Time to Macrophage Activation Syndrome (MAS) laboratory remission | From Index date up to 26 weeks
  Time to normalization for all key laboratory values
Time to partial MAS laboratory remission | From Index date up to 26 weeks
  Time to normalization for at least 3 key laboratory values
Time to tapering of Glucocorticoids (GCs) | from index date to the last of 7 consecutive days
  From index date to the last of 7 consecutive days receiving ≤1 mg/kg/day of prednisone (PDN).
Number of recurrent MAS episodes | through study completion
  Occurring any time after the end of the data collection period for the index MAS episode
Administration of organ support care | from the index date until either the end of hospitalization or 26 weeks, whichever occurs later
  Proportion of patients receiving hemodialysis, assisted ventilation, cardiac support, or inotropic drugs
Characteristics of MAS treatment | for MAS episodes occurring during the data collection period
  description of treatment patterns of MAS-related treatments for both index and recurrent MAS episodes.
Clinical signs | At index date and 8 weeks after index date or at the earliest time this data becomes available between 8 and 12 weeks
  No of MAS symptoms (Fever, Skin rash, Hemorrhagic manifestations, Evidence of CNS involvement) present

SECONDARY OUTCOMES:
Time to hospital discharge | Up to 26 weeks
  Defined as time from the index date to discharge from the hospital
Time to intensive care unit (ICU) discharge | Up to 26 weeks
  For patients who are admitted to the ICU during the index MAS episode, this is defined as time from index date or ICU admission (whichever comes later) to ICU discharge
Duration of Clinical Response | Until week 26
  defined as the time (in days) from the date of first documented MAS laboratory remission until the date of first documented occurrence of a new MAS episode as per investigator's assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Ullman, MD, Study Director — Swedish Orphan Biovitrum AG Riehenring 182, 4058 Basel, Switzerland
Locations (11):
- United States (4):
  - Swedish Orphan Biovitrum Research Site, Los Angeles, California
  - Swedish Orphan Biovitrum Research Site, Atlanta, Georgia
  - Swedish Orphan Biovitrum Research Site, Cincinnati, Ohio
  - Swedish Orphan Biovitrum Research Site, Philadelphia, Pennsylvania
- Swedish Orphan Biovitrum Research Site, Calgary, Canada
- Swedish Orphan Biovitrum Research Site, Paris, France
- Swedish Orphan Biovitrum Research Site, Heidelberg, Germany
- Italy (2):
  - Swedish Orphan Biovitrum Research Site, Milan
  - Swedish Orphan Biovitrum Research Site, Rome
- Swedish Orphan Biovitrum Research Site, Utrecht, Netherlands
- Swedish Orphan Biovitrum Research Site, Barcelona, Spain